CLINICAL TRIAL: NCT07218549
Title: Evaluation of the Safety and Effects of Psychoactive Substances in People With Past Opioid Use
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Christopher D. Verrico (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Christopher D. Verrico, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H-56391
Record Dates: First submitted 2025-09-18; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use; Substance Use Disorders; Opioid Analgesia
Keywords: Opioid Use; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: 6-way crossover study to determine the abuse potential of kratom relative to oxycodone and placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment Sequence A (Placebo Comparator): Placebo: A single dose of placebo to match kratom (over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Placebo
- Treatment Sequence B (Active Comparator): Active Control: A single 20 mg dose of oxycodone (1 X 20 mg tablet over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Oxycodone HCl
- Treatment Sequence C (Active Comparator): Active Control: A single 40 mg dose of oxycodone (2 X 20 mg tablets over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Oxycodone HCl
- Treatment Sequence D (Experimental): Kratom: A single 8 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Kratom 8
- Treatment Sequence E (Experimental): Kratom: A single 12 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Kratom 12g
- Treatment Sequence F (Experimental): Kratom: A single 16 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Interventions: Drug: Kratom 16g

INTERVENTIONS:
Drug: Placebo — Placebo: A single dose of placebo to match kratom (over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence A
Drug: Oxycodone HCl — Active Control: A single 20 mg dose of oxycodone (1 X 20 mg tablet over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence B
Drug: Oxycodone HCl — Active Control: A single 40 mg dose of oxycodone (2 X 20 mg tablets over-encapsulated placebo in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence C
Drug: Kratom 8 — Kratom: A single 8 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence D
Drug: Kratom 12g — Kratom: A single 12 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence E
Drug: Kratom 16g — Kratom: A single 16 g dose of kratom (in 32 opaque 00 capsules) will be administered orally.
  Arms: Treatment Sequence F

SUMMARY:
This research study intends to evaluate the safety and tolerability of commonly used drugs or substances on recreational drug users with experience of using any of the following: heroin, oxycodone, kratom, morphine, cocaine, fentanyl, PCP, LSD, cocaine, etc. Another objective of the study is to evaluate the pharmacokinetics and pharmacodynamics of the drugs administered to you. Pharmacokinetics is the study of how a drug is absorbed into the blood, circulated, broken down, and eventually eliminated by the body. Pharmacodynamics is the study of the drug's effects on the body, including how it makes you feel.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking, 18- to 55-year-old males or females.
2. Female subjects must have a negative serum pregnancy test at time of screening and negative urine pregnancy test upon admission. In addition, female subjects must meet one of the following conditions:

   * Is a woman of non-childbearing potential defined as no menses for at least 12 months with status confirmed by FSH and estradiol levels at screening or surgically sterile at screening visit OR
   * Is a woman of childbearing potential and using a contraceptive method that is highly effective, with a failure rate of <1%, from Screening until 9 months after receiving the study medication. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the dose of study intervention.
3. Male subjects must agree to the following from Day 1 until 9 months after receiving the study medication:

   • Not donate fresh unwashed semen

   Plus, either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
   * Use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
   * Use a male condom when engaging in any activity that allows for passage of ejaculate to another person
4. Physically healthy, as determined by a clinical interview with a physician, laboratory tests (urinalysis, blood chemistry, 12-lead ECG), physical examination, and self-reported medical history.
5. No current or past diagnosis of severe mental illness, as determined by a clinical interview.
6. Clinical laboratory test results (CMP, CBC, etc.) must be within the normal reference range or with acceptable deviations that are judged to be not clinically significant by a study physician.
7. Have a history of self-reported recreational opioid use as defined by at least 10 times in the past year and at least once in the 12 weeks before screening.
8. Able and willing to give signed informed consent, reliable, and willing to make themselves available for the study's duration and follow study procedures.
9. Agree not to consume any recreational drugs during the study (THC is excluded).
10. Able to perform study procedures as determined by clinical judgment.
11. Able to meet eligibility requirements of the Qualification Phase (i.e., drug discrimination) and Naloxone Challenges.

Exclusion Criteria:

1. Seeking treatment for a substance or alcohol use disorder as determined by self-report during the intake interview.
2. Current or past diagnosis of opioid use disorder or other substance use disorder (SUD) within the past year, excluding THC and nicotine-containing products. With regard to marijuana/THC, an individual must be able to tolerate 48 hours of abstinence from marijuana/THC products.
3. History of opioid overdose.
4. Using medication or supplements that might interact with kratom or oxycodone as determined by self-report during intake interview.
5. Treatment with any investigational drug during the last 30 days.
6. Participants on parole or probation.
7. Currently pregnant or trying to conceive or currently lactating as determined by blood pregnancy testing at screening, urine pregnancy testing at admission, and self-reporting during interview and study visits.
8. Current or recent history of significant violent or suicidal behavior or suicidal/homicidal risk as determined by the C-SSRS.
9. Sensitivity, allergy, or contraindications/allergies to kratom, opioids, or similar compounds.
10. Use prescription or nonprescription drugs and dietary supplements within seven days or five half-lives (whichever is longer) that, in the opinion of the study clinician may interfere with the investigational product.
11. Positive urine drug screen (UDS) for substances of abuse at each admission in the Qualification and Treatment phases, excluding tetrahydrocannabinol (THC). If a participant presents with a positive UDS excluding THC at any admission or any visit, the investigator, at their discretion, may reschedule a repeat of UDS until the UDS is negative, excluding THC, before the participant is permitted to participate in any phase of the study.
12. Positive alcohol breathalyzer test at each admission in the Qualification and Treatment Phase.
13. History of sensitivity to heparin or heparin-induced thrombocytopenia.
14. Has not donated blood or plasma within the last six weeks.
15. Has a history of increased intracranial pressure or brain tumors.
16. Has gastrointestinal obstruction, including paralytic ileus.
17. Has a history of seizure disorders.
18. Has a chronic obstructive pulmonary disease or cor pulmonale.
19. Has a history of anemia or any other significant hematologic disorder.
20. Has a condition or abnormality that, in the opinion of the PI or Study Physician, would compromise the safety of the patient or the quality of the data.
21. Has a major surgery planned within the next 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Drug Liking Visual Analog Scale | From Treatment Week 1 to Treatment Week 8
  The primary endpoint of this study will be maximum (peak) effect (Emax) over 24 hours for Drug Liking ("at this moment"), assessed on a bipolar (0 to 100 points) visual analog scale (VAS).

SECONDARY OUTCOMES:
Overall Drug Liking Visual Analog Scale | From Treatment Week 1 to Treatment Week 8
  Overall drug liking of the study products will be assessed 12 and 24 hours following each dose in the Treatment phase. VAS assessments will be scored on a 100-point scale, where a rating of "0" reflects the complete absence of a subjective effect while a rating of "100" reflects the maximum presence of a subjective effect.
Take Drug Again Visual Analog Scale | From Treatment Week 1 to Treatment Week 8
  Take Drug Again will be assessed 12 and 24 hours following each dose in the Treatment phase. VAS assessments will be scored on a 100-point scale, where a rating of "0" reflects the complete absence of a subjective effect while a rating of "100" reflects the maximum presence of a subjective effect.
Pharmacokinetic (PK)- maximum observed concentration (Cmax) | Treatment Week 1 to Treatment Week 8
  Pharmacokinetic parameters of kratom alkaloids include maximum observed concentration (Cmax).
Safety- Adverse Events | Treatment Week 1 to Treatment Week 8
  Endpoints will include a summary of the incidence of adverse events (AEs), serious adverse events (SAEs), as well as descriptive summary and statistics of the safety parameters.
Pharmacokinetic (PK)- time of last measurable observed concentration (Tlast) | Treatment Week 1 to Treatment Week 8
  Pharmacokinetic parameters of kratom alkaloids include time of last measurable observed concentration (Tlast).
Pharmacokinetic (PK)- area under the curve from time 0 to the last measurable observed concentration (AUC0-T) | Treatment Week 1 to Treatment Week 8
  Pharmacokinetic parameters of kratom alkaloids include the area under the curve from time 0 to the last measurable observed concentration (AUC0-T).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Verrico, PhD Pharmacology, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No